CLINICAL TRIAL: NCT06392646
Title: The Effect of a Postoperative Education Programme Based on Swanson's Theory of Caring on the Self-management Behavioural Competence of Elderly Enterostomal Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuxi No. 2 People's Hospital (Other)
Responsible Party: Principal Investigator, Xue Yan, nurse, Wuxi No. 2 People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Wuxi2PH
Record Dates: First submitted 2024-04-24; First posted 2024-04-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Enterostomy; Elderly; Self-management; Education
Keywords: Enterostomy; elderly; self-management; education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine care (No Intervention): Taking routine care measures
- self-management education program (Experimental): Intervention in accordance with the constructed self-management education program
  Interventions: Behavioral: self-management education program

INTERVENTIONS:
Behavioral: self-management education program — Intervention through a self-management education program constructed through evidence summarization and expert correspondence.
  Arms: self-management education program

SUMMARY:
The purpose of this intervention study was to understand the impact of a self-management education program on self-management skills, quality of life, and caregiver burden in older patients with enterostomies. It aims to answer the main question of whether a self-management education program can improve self-management skills, quality of life, and reduce family caregiver burden in elderly patients with enterostomies.

ELIGIBILITY:
Inclusion Criteria:

* age ≥60 years
* first enterostomy surgery
* informed consent to voluntarily participate in this study.

Exclusion Criteria:

* verbal communication disorder; cognitive dysfunction or history of mental illness;
* visual and manual mobility impairment unable to perform stoma care operations.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
self-management | during hospitalization, approximately 5 days and post-discharge, 1month
  Self-management behavior questionnaire for patients with enterostomies. The questionnaire has a total score of 40-200, with higher scores being associated with better stoma self-management behaviours.
the quality of life | during hospitalization, approximately 5 days and post-discharge, 1month
  City of Hope Quality of Life-ostomy Questionaire, COH-QOL-OQ. The scale has a total score of 0-320, with higher scores being associated with higher quality of life.
Caregiver burden | during hospitalization, approximately 5 days and post-discharge, 1month
  Zarit Burden Interview,ZBI. The scale is scored on a total scale of 0-88, with the higher the score, the higher the burden on the carer.

CONTACTS AND LOCATIONS:
Locations (1):
- Yan Xue, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No